CLINICAL TRIAL: NCT06933550
Title: FFG PREMEDICAL (Clinical Investigation of a Medical Device According to MDR Article 82, Para.1 and Austrian Law §13 Para. 3 MPG, BGBI. I No. 122/2021 - Study Without Influence on Diagnostics/Therapy)
Brief Title: PREMEDICAL is a Clinical Investigation Aiming to Create a Data Basis That Can be Used to Enrich Information Collected in the Course of the Classic Patient Journey. Patients in the Emergency Department Will be Asked to Answer Patient-related and Symptom-oriented Questions. Minimum Age is 18 Years
Status: Not yet recruiting | Type: Observational
Sponsor: XUND Solutions GmbH (Industry)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 892459; 102478757 (Other: BASG/AGES Institute Surveillance)
Record Dates: First submitted 2025-04-08; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Emergency Department Triage
Keywords: XUND; emergency department; symptom check; patient journey
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
The goal of this clinical investigation is to create a new type of data basis that can be used to enrich information collected in the course of the classic patient journey, such as medical history forms and discharge letters. Therefore, it is planned to collect new, patient-related and symptom-oriented data on site and directly from patients in the emergency department (female/male; at least 18 years old).

The main question it aims to answer is:

- Can a detailed medical history with additional enriched information from XUND improve the quality of outpatient care?

Selected patients in the waiting area of the emergency department will record their symptoms on a tablet and answer the questions asked about their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a signed informed consent form;
* signed consent and admission to the emergency department of the emergency medicine clinic
* Triage category 3, 4 or 5 based on the triage procedure according to the Manchester triage system used in Austria
* the physical and mental ability to operate the tablet and answer the questions
* 18 years of age or older;
* knowledge of the German language.

Exclusion Criteria:

* not meeting all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German speaking, at least 18 years old, all gender patients in the emergency department (triage category 3, 4, or 5).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
XUND Symptom Checker | through investigation completion, an average of 1 year
  The fundamental element of the proposed project is the aggregation of novel, patient-related and symptom-oriented data on-site and directly from patients in the emergency department. The objective of this study is to establish a novel type of data basis, with the potential to enhance the information collected during the conventional patient journey, including medical history forms and discharge letters. XUND's Symptom Check, which has been certified as a class IIa medical device, will be used to collect the data. Selected patients in the emergency waiting area record their symptoms on a tablet and answer the questions asked. The Symptom Check is powered by an AI-driven medical knowledge base of 520+ conditions and 21,000+ symptom variants.

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Peter Kamolz, Univ. Prof. Dr., Principal Investigator — Medizinische Universität Graz, Universitätsklinik für Chirurgie
Locations (1):
- Medical University of Graz, Graz, Austria